CLINICAL TRIAL: NCT04736485
Title: Perioperative Treatment in Resectable Gastric Cancer With Spartalizumab (PDR001) in Combination With Fluorouracil, Leucovorin, Oxaliplatin, and Docetaxel (FLOT): A Phase II Study (GASPAR)
Brief Title: Perioperative Treatment in Resectable Gastric Cancer With Spartalizumab (PDR001) in Combination With Fluorouracil, Leucovorin, Oxaliplatin, and Docetaxel (FLOT)
Acronym: GASPAR
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Centre Francois Baclesse (Other)
Collaborators: National Cancer Institute, France (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020-004497-21
Record Dates: First submitted 2021-01-26; First posted 2021-02-03 (Actual); Last update posted 2022-12-23 (Actual); Status verified 2022-12

CONDITIONS: Gastric Cancer by AJCC V8 Stage; Resectable Carcinoma
Keywords: perioperative; spartalizumab; PDR001; Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- FLOT regimen plus Spartalizumab (Experimental): Standard FLOT regimen
  * Docetaxel 50 mg/m² IV infusion on D1
  * Oxaliplatine 85 mg/m² IV infusion on D1
  * Leucovorin 200 mg/m² IV infusion on D1
  * Fluorouracile 2600 mg/m² 24 h IV infusion on D1
  with Spartalizumab PDR001 Patients will received the fixed dose of 400 mg per IV infusion on D1 every four weeks (q4w) for 2 pre-operative cycles (8 weeks) and 2 post-operative cycles (8 weeks)
  Interventions: Drug: perioperative treatment

INTERVENTIONS:
Drug: perioperative treatment — FLOT + Spartalizumab

SUMMARY:
Multicenter, open-label, non randomized, phase 2 trial in resectable gastric or gastroesophageal junction adenocarcinoma: Perioperative Treatment by Spartalizumab (PDR001) in Combination with fluorouracil, leucovorin, oxaliplatin, and docetaxel (FLOT)

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Untreated localized gastric or GEJ adenocarcinoma considered resectable (clinical stage ≥cT2 and/or cN+ and no metastasis)
* Histologically confirmed adenocarcinoma
* ECOG performance status score of 0 or 1
* Tumor tissue must be provided for biomarker analyses (fresh or archival with an FFPE tissue block)
* All subjects must consent to allow the acquisition of blood samples for performance of correlative studies
* Screening laboratory values must meet the following criteria:

  * WBC ≥ 2000/ mm³
  * Neutrophils ≥ 1500/ mm³
  * Platelets ≥ 100 000/ mm³
  * Hemoglobin ≥ 9.0 g/dL
  * Bilirubin ≤ 1.5 x ULN, AST and ALT ≤ 3 x ULN
  * Measured or calculated creatinine ≥ 50 ml/min clearance (CrCl) (using the Cockcroft-Gault formula)
  * Potassium ≥ LLN
  * Magnesium ≥ LLN
  * Calcium ≥ LLN
* Female subject of childbearing potential must have a negative urine or serum pregnancy test within 72h before study start
* Subject in reproductive age must be willing to use adequate contraception during the study and at least 9 months in men and 12 months in women after the last dose of investigational drug. In addition, given the toxicities observed on the male reproductive system, a conservation of gametes will be proposed for men, as usually in routine practice
* Subject affiliated to a social security regimen
* Patient has signed informed consents obtained before any trial related activities and according to local guidelines

Exclusion Criteria:

Subject with any distant metastasis

* Subject with no recovering from the effects of major surgery or significant traumatic injury within 14 days before inclusion
* Documented significant cardiovascular disease within the past 6 months before the first dose of study treatment, including: history of congestive heart failure (defined as NYHA III or IV), myocardial infarction, unstable angina, coronary angioplasty, coronary stenting, coronary artery bypass graft, cerebrovascular accident or hypertensive crisis
* History of anterior organ transplant, including stem cell allograft
* Pneumonitis or interstitial lung disease
* History of other malignancy within the previous 3 years (except for appropriately treated in-situ cervix carcinoma and non-melanoma skin carcinoma)
* Subject with active, known, or suspected autoimmune disease
* Subject with a condition requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalent) or other immunosuppressive medications within 14 days of start of study treatment GASPAR Protocol - EUDRACT number: 2020-004497-21 - version 1.3 / 2021-01-18 Page 8 sur 44
* Known history of HIV or HBV infection
* Known active HCV infection
* Known history of active tuberculosis
* Vaccination with live vaccine within 30 days before the first dose of study treatment
* Prior treatment with an anti-PD-1, anti-PD-L1, anti-PD-L2 or any other antibody or drug specifically targeting T-cell co-stimulation or checkpoint pathways
* Recent or concomitant treatment with brivudine (herpes virostatic)
* Prior anticancer therapy for the current malignancy
* Known hypersensitivity to any of the study drugs or their excipients
* Chronic inflammable gastro-intestinal disease
* Uracilemia ≥ 16 ng/ml
* QT/QTc > 450 msec for men and > 470 msec for women
* Peripheral neuropathy ≥ Grade II
* Uncontrolled diabetes
* Active infection requiring systemic therapy
* Participation in another therapeutic clinical study
* Patient deprived of liberty or placed under the authority of a tutor
* Patient assessed by the investigator to be unable or unwilling to comply with the requirements of the protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Estimated)
Dates: Start 2021-06-28 (Actual); Primary Completion 2024-03 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Pathologic response after pre-operative treatment | At surgery, an average 3 months after treatment initiation
  Proportion of patients with pCR (pathologic complete response) in the primary tumour defined as: no tumour residue found in the tissue collected during the surgery evaluated by the pathologist

SECONDARY OUTCOMES:
Evaluate the impact of perioperative treatment on disease-free survival | Through study completion, an average of 5 follow-up year
  Disease-free survival (DFS) defined as time between inclusion and first disease progression
Evaluate the impact of perioperative treatment on overall survival | Up to death
  Overall survival (OS) defined as the time between inclusion and death whatever cause;
The correlation between pathologic Complete response and survival outcomes (disease-free and overall survival) | At surgery, an average 3 months after treatment initiation
  Proportion of patients with margin-free resection (R0), defined as a microscopically margin-negative resection, in which no gross or microscopic tumor remains in the primary tumor bed
Treatment-Related Adverse Events | Toxicities occurring up to 1 month after the end of treatment
  Type, grade and number of Adverse Events as Assessed by CTCAE v5.0

CONTACTS AND LOCATIONS:
Locations (13):
- France (13):
  - CHU Besançon, Besançon
  - Centre François Baclesse, Caen
  - Centre Georges Francois Leclerc, Dijon
  - Chru Lille, Lille
  - APHM Marseille, Marseille
  - Institut Régional Cancer, Montpellier
  - APHP St Louis, Paris
  - Institut Mutualiste Montsouris, Paris
  - CHU Poitiers, Poitiers
  - CHU Robert Debré, Reims
  - Centre Eugène Marquis, Rennes
  - ICO St Herblain, Saint-Herblain
  - CH St Malo, St-Malo

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Dos Santos M, Lequesne J, Piessen G, Leconte A, Guimbaud R, Pernot S, Bouche O, Hiret S, Soularue E, Tougeron D, Dahan L, Le Sourd S, Borg C, Samalin E, Corbinais S, Parzy A, Guilloit JM, Varatharajah S, Brachet PE, Dorbeau M, Galais MP, Desgrippes R, Clarisse B. Perioperative treatment in resectable gastric cancer with spartalizumab in combination with fluorouracil, leucovorin, oxaliplatin and docetaxel (FLOT): Results from the GASPAR phase 2 study. Eur J Cancer. 2026 Jan 30;236:116258. doi: 10.1016/j.ejca.2026.116258. Online ahead of print. PMID 41653501
- [Derived] Dos Santos M, Lequesne J, Leconte A, Corbinais S, Parzy A, Guilloit JM, Varatharajah S, Brachet PE, Dorbeau M, Vaur D, Weiswald LB, Poulain L, Le Gallic C, Castera-Tellier M, Galais MP, Clarisse B. Perioperative treatment in resectable gastric cancer with spartalizumab in combination with fluorouracil, leucovorin, oxaliplatin and docetaxel (FLOT): a phase II study (GASPAR). BMC Cancer. 2022 May 12;22(1):537. doi: 10.1186/s12885-022-09623-z. PMID 35549674